CLINICAL TRIAL: NCT06478940
Title: Clinical and Radiographic Evaluation of 3Mixtatin Versus MTA Used as Pulpotomy Agents in Vital Primary Molars: A Randomized Clinical Trial
Brief Title: 3Mixtatin and MTA Vital Pulpotomy in Primary Molars
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sally Ahmed Kotb, doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3Mixtatin and MTA pulpotomy
Record Dates: First submitted 2024-06-23; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Pulp Disease, Dental; Deciduous Teeth
Keywords: pulpotomy - vital pulp therapy; primary molars- baby teeth
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTA pulpotomy (Active Comparator): pulpotomy with MTA applied in the vital pulp therapy
  Interventions: Drug: MTA pulpotomy
- 3 Mixtatin pulpotomy (Experimental): pulpotomy with 3 mixtatin (triple antibiotic paste of (Metronidazole, cefixime, and Ciprofloxacin mixed with simvastatin ) applied in the vital pulp therapy
  Interventions: Drug: 3 mixtatin pulpotomy

INTERVENTIONS:
Drug: 3 mixtatin pulpotomy — pulp treatment with applying 3mixture of antibiotic (Metronidazole, cefixime, and Ciprofloxacin) along with simvastatin
  Arms: 3 Mixtatin pulpotomy
Drug: MTA pulpotomy — pulp treatment with applying MTA
  Arms: MTA pulpotomy

SUMMARY:
The aim of the study is to evaluate clinical and radiographic success of using 3Mixtain versus mineral trioxide aggregate in pulpotomy of deeply carious Primary molars.

DETAILED DESCRIPTION:
Due to the complexity of the root canal microbiome, it is doubtful that they can be treated properly with a single antibiotic. Accordingly, a combination of multiple antibiotics seemed to be essential to diminish different types of pathogenic bacteria. Recently, a combination of three antibiotics (Metronidazole, cefixime, and Ciprofloxacin) along with Statins (new bio-inductive materials in regenerative dentistry) has shown promising results in primary teeth pulp therapy.

Statin components have an anti-inflammatory impact on pulp tissue by lowering the amount of interleukin-6 and interleukin-8. They also decrease osteoclastic processes and strengthen osteoblastic processes. Thus, they promote bone regeneration and dentin formation by enhancing odontoblastic activity. Several studies have shown a clinical and radiographic success rate of 3Mixtatin with inconsistent results. Some randomized controlled Trials (RCTs) showed that MTA had a comparable result with 3Mixtatin, while others reported that 3Mixtatin might be an alternative for MTA due to its higher overall success rate. 3Mixtatin is considered as a novel material with successful outcomes. Owing to limited availability of data in researches and in order to reach a conclusive results our study aims to evaluate clinical and radiographic success of using 3Mixtain versus mineral trioxide aggregate in pulpotomy of deeply carious Primary molars .

ELIGIBILITY:
Inclusion Criteria:

* • Children 4-8 years old

  * Vital deeply carious primary molars.
  * No history of spontaneous pain, pathologic mobility, draining sinus tract, redness or swelling of the vestibule.
  * Normal gingival and periodontal condition, with no sensitivity to vestibular palpation, and no pain on percussion test.
  * Patient and parent showing cooperation and compliance.

Exclusion Criteria:

* • Uncooperative children to avoid time waste and attrition bias.

  * Unrestorable molars
  * Sign of radiolucency in periapical or furcation area
  * Widening of PDL space or loss of lamina dura continuity
  * Evidence of internal/external pathologic root resorption
  * During operative procedure, when hemorrhage control is not achievable after pulpotomy.
  * Children with systemic disease as some systemic diseases may have effect on the outcome.
  * Unable to attend follow-up visits to avoid attrition bias by decreasing number of drop off cases.
  * Refusal of participation as the parent of child has the authority of participation.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success Clinical success clinical success | 1 week , 3 months , 6 months , 9 months and 12 months
  absence of postoperative pain,Absence of pain on percussion,Absence of Swelling and Absence of Sinus or fistula

SECONDARY OUTCOMES:
Radiographic success radiographic success | 3 months , 6 months , 12 months
  Absence of any adverse radiographic findings (Periodontal membrane space widening, bone resorption, pulp stones, internal or external root resorption )

CONTACTS AND LOCATIONS:
Overall Officials: Randa y Abd Al Gawad, professor, Study Director — Professor of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University; Yasmin M Yousry, Associate professor, Study Chair — Assistant Professor of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University

REFERENCES:
- [Background] Almarji W, Laflouf M, Tolibah YA. Evaluation of the modified 3Mix-Simvastatin combination in non-instrumental endodontic therapy of necrotic primary molars: A two-arm randomized controlled trial. Clin Exp Dent Res. 2024 Apr;10(2):e860. doi: 10.1002/cre2.860. PMID 38433296
- [Background] Zarabadi MS, Firoozi P, Basir Shabestari S, Maleki A, Nazemi Salman B. 3Mixtatin versus MTA in pulp therapy of primary teeth: a systematic review and meta-analysis of current randomized controlled trials. Evid Based Dent. 2024 Jun;25(2):111-112. doi: 10.1038/s41432-024-00987-8. Epub 2024 Mar 6. PMID 38448571
- [Background] Mushtaq A, Nangia T, Goswami M. Comparative Evaluation of the Treatment Outcomes of Pulpotomy in Primary Molars Using Mineral Trioxide Aggregate and 3Mixtatin: A Randomized Clinical Trial. Int J Clin Pediatr Dent. 2023 Nov-Dec;16(6):810-815. doi: 10.5005/jp-journals-10005-2720. PMID 38344366
- [Background] Chak RK, Singh RK, Mutyala J, Killi NK. Clinical Radiographic Evaluation of 3Mixtatin and MTA in Primary Teeth Pulpotomies: A Randomized Controlled. Int J Clin Pediatr Dent. 2022;15(Suppl 1):S80-S86. doi: 10.5005/jp-journals-10005-2216. PMID 35645497
- [Background] Aminabadi NA, Huang B, Samiei M, Agheli S, Jamali Z, Shirazi S. A Randomized Trial Using 3Mixtatin Compared to MTA in Primary Molars with Inflammatory Root Resorption: A Novel Endodontic Biomaterial. J Clin Pediatr Dent. 2016;40(2):95-102. doi: 10.17796/1053-4628-40.2.95. PMID 26950808
- [Background] Asl Aminabadi N, Satrab S, Najafpour E, Samiei M, Jamali Z, Shirazi S. A randomized trial of direct pulp capping in primary molars using MTA compared to 3Mixtatin: a novel pulp capping biomaterial. Int J Paediatr Dent. 2016 Jul;26(4):281-90. doi: 10.1111/ipd.12196. Epub 2015 Sep 15. PMID 26370520
- [Background] Goel N, Kumar A, Singhal R, Jha S, Namdev R, Rani R. Comparative Evaluation of Chlorhexidine Polymer Scaffold, 3Mixtatin, and Formocresol for Vital Primary Pulp Therapy: A Randomized 6-month Clinical Study. Int J Clin Pediatr Dent. 2023 May-Jun;16(3):478-482. doi: 10.5005/jp-journals-10005-2615. PMID 37496952
- [Background] Jamali Z, Alavi V, Najafpour E, Aminabadi NA, Shirazi S. Randomized Controlled Trial of Pulpotomy in Primary Molars using MTA and Formocresol Compared to 3Mixtatin: A Novel Biomaterial. J Clin Pediatr Dent. 2018;42(5):361-366. doi: 10.17796/1053-4625-42.5.7. Epub 2018 May 15. PMID 29763354